CLINICAL TRIAL: NCT05562921
Title: A Pilot Study of Hypertension Management Using Remote Patient Monitoring- Extended Follow Up Using Matched Cohort Design
Brief Title: Hypertension Management Using Remote Patient Monitoring
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Omron Healthcare Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Stephen Persell, MD, MPH, Professor, Northwestern University
Other Study IDs: STU00213093-3
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case
  Interventions: Behavioral: Cases-remote patient monitoring prescribed
- Control
  Interventions: Behavioral: Controls-ususal care

INTERVENTIONS:
Behavioral: Controls-ususal care — Controls: patients who did not receive remote patient monitoring for blood pressure prescribed during routine care delivery, with multivariable matching to cases
  Groups: Control
Behavioral: Cases-remote patient monitoring prescribed — Cases: patients prescribed remote patient monitoring for blood pressure during routing care delivery
  Groups: Case

SUMMARY:
A longer-term follow-up of patients with remote patient monitoring ordered from the initial six pilot primary care clinics (from the prior study periods: Study 1 and Study 2) will be performed and compared to a cohort of patients without RPM orders, matched on clinical and demographic characteristics, from the same six pilot primary care clinics, to serve as contemporary controls.

ELIGIBILITY:
Inclusion Criteria Cases Patients from any of 6 primary care sites that participated in remote monitoring pilots who had remote patient monitoring (RPM) ordered by a primary care clinician between November 18, 2018 and August 14, 2021

-

Exclusion Criteria:

* Patients whose RPM ordered by non-primary care clinics

Matching cohort Inclusion

* Patients from the six pilot clinics AND
* Meet the matching criteria Exclusion
* Patients with any RPM order between between November 18, 2018 and August 14, 2021

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Case population includes patients with RPM for blood pressure ordered from the six pilot primary care clinics between November 18, 2018 and August 14, 2021, are 65 to 85 years old, and have Medicare insurance.
  Control population are patients selected from the same practices using propensity score matching who were not prescribed RPM for blood pressure.
Sampling Method: Non-Probability Sample
Enrollment: 1440 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Controlling High Blood Pressure (NQF 0018) | 18 months
  Proportion of patients who satisfy the performance measure Controlling High Blood Pressure (NQF 0018), last BP done within 1 year and is less than 140/90 mm Hg
Controlling High Blood Pressure (NQF 0018) | 15 months
  Proportion of patients who satisfy the performance measure Controlling High Blood Pressure (NQF 0018), last BP done within 1 year and is less than 140/90 mm Hg
Controlling High Blood Pressure (NQF 0018) | 12 months
  Proportion of patients who satisfy the performance measure Controlling High Blood Pressure (NQF 0018), last BP done within 1 year and is less than 140/90 mm Hg

SECONDARY OUTCOMES:
Antihypertensive medication intensification | 18 months
  Count of antihypertensive medication drug classes added or increased during the time frame minus the number decreased or discontinued
Antihypertensive medication intensification | 15 months
  Count of antihypertensive medication drug classes added or increased during the time frame minus the number decreased or discontinued
Antihypertensive medication intensification | 12 months
  Count of antihypertensive medication drug classes added or increased during the time frame minus the number decreased or discontinued

OTHER OUTCOMES:
Mean SBP at most recent office visit | 18 months
  Mean SBP at most recent office visit
Mean SBP at most recent office visit | 15 months
  Mean SBP at most recent office visit
Mean SBP at most recent office visit | 12 months
  Mean SBP at most recent office visit
Mean SBP on most recent measurement date (office or out of office) | 18 months
  Mean SBP on most recent measurement date (office or out of office)
Mean SBP on most recent measurement date (office or out of office) | 15 months
  Mean SBP on most recent measurement date (office or out of office)
Mean SBP on most recent measurement date (office or out of office) | 12 months
  Mean SBP on most recent measurement date (office or out of office)
Ambulatory care utilization--office visits | 18 months
  Count of primary care office visits during time frame
Ambulatory care utilization--telephone calls | 18 months
  Count of primary care telephone encounters during time frame
Ambulatory care utilization--patient portal messages | 18 months
  Count of primary care patient portal encounters during time frame
Proportion of patients with an increase in serum creatinine of ≥30% | 18 months
  Proportion of patients with an increase in serum creatinine of ≥30%

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Persell, MD/MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petito LC, Anthony L, Peprah Y, Lee JY, Li J, Sato H, Persell SD. Blood pressure outcomes at 12 months in primary care patients prescribed remote physiological monitoring for hypertension: a prospective cohort study. J Hum Hypertens. 2023 Dec;37(12):1091-1097. doi: 10.1038/s41371-023-00850-w. Epub 2023 Jul 21. PMID 37479812